CLINICAL TRIAL: NCT03923530
Title: Pressure Assessment to Improve Outcomes After TAVR: a Registry
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: Malcom Randall VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony Bavry, Director of Cardiovascular Catheterization Laboratory, North Florida Foundation for Research and Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201901097
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Aortic Stenosis, Calcific; Quality of Life; Heart Failure With Preserved Ejection Fraction
Keywords: TAVR; KCCQ; Aortic stenosis; Diastolic dysfunction; Invasive hemodynamic assessment
MeSH Terms: conditions — Hypertension; Aortic Valve, Calcification of; Aortic Valve Stenosis | interventions — Eplerenone

STUDY DESIGN:
Intervention Model Description: Enroll subjects who underwent TAVR and had documentation of abnormal invasive cardiac hemodynamics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eplerenone (Experimental): Eplerenone 50 mg daily, administered orally for 8 weeks.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 50 mg daily
  Other Names: Inspra

SUMMARY:
At the Malcom Randall Veterans Affairs Medical Center (MRVAMC), invasive cardiac pressures are routinely recorded after transcatheter aortic valve replacement (TAVR) procedures. Our research has disclosed that patients with abnormal hemodynamics (narrow aortic to ventricular end-diastolic pressure difference, indexed to heart rate) suffer from high long-term mortality, compared with patients with normal hemodynamics.This hemodynamic value can be referred to as the aortoventricular index (AVi). Hypertension and diastolic dysfunction are highly co-morbid conditions among these patients. The selective aldosterone receptor antagonist eplerenone (Inspra) is approved for use in the treatment of hypertension. Research also supports that eplerenone may be able to improve diastolic function.

This prospective study is interested in determining 1) the tolerability of eplerenone, and 2) feasibility of administering the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) among subject with abnormal cardiac hemodynamics after TAVR. This study will set the stage for a pilot randomized trial to evaluate eplerenone versus placebo among patients with abnormal hemodynamics after TAVR.

DETAILED DESCRIPTION:
Our research has disclosed that patients who have abnormal invasive cardiac hemodynamics (narrow aortic to ventricular end-diastolic pressure difference, indexed to heart rate) after TAVR suffer from poor long-term survival. This hemodynamic value can be referred to as the aortoventricular index (AVi). In a single center observational study, the 2-year mortality rate for patient with a value ≥0.6 mm Hg/bpm was 25% compared with 36% for patients with a value <0.6 mm Hg/bpm. An abnormal AVi was an independent predictor for poor survival. Hypertension and diastolic dysfunction are 2 highly co-morbid conditions among these patients. Currently, there is lack of appreciation that pressure measurements obtained at the time of TAVR can provide long-term prognostic value. There is also a lack of understanding on how to improve outcomes and quality of life among such patients.

Eplerenone is a selective aldosterone receptor antagonist approved for use for treatment of hypertension. Animal studies have shown that aldosterone receptor antagonists can decrease interstitial myocardial fibrosis. The non-selective aldosterone receptor antagonist, spironolactone 25 mg daily compared with placebo was shown to improve diastolic function, as assessed by echocardiography, among 28 elderly subjects. A meta-analysis of eleven studies in 942 subjects found that aldosterone receptor antagonists improve diastolic function and markers of cardiac fibrosis without significant changes to left ventricular mass or dimensions. In a randomized controlled trial, eplerenone was found to be safely tolerated among asymptomatic patients with moderate to severe aortic stenosis.

ELIGIBILITY:
1. Enroll 10 subjects with hypertension and abnormal hemodynamics after TAVR.
2. This is a greater than minimal risk study.

   1. Inclusion criteria:

      * TAVR procedure performed at the Malcom Randall VA Medical Center within the last 2 years.
      * Intracardiac pressures recorded 5 to 10 minutes after TAVR and AVi < 0.6 mm Hg/bpm.
      * History of hypertension, taking anti-hypertensive medications, or recent systolic blood pressure ≥130 mm Hg.
   2. Exclusion criteria:

      * Serum potassium >5.5 mEq/L at initiation.
      * Concomitant administration of strong CYP3A inhibitor (i.e. ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, and nelfinavir).
      * Type 2 diabetes with microalbuminuria.
      * Serum creatinine >2.0 for men and >1.8 for women.
      * Creatinine clearance <50 cc/min.
      * Concomitant administration of potassium supplements or potassium-sparing diuretics.
3. Subjects who are eligible to participate and signed an informed consent will be given eplerenone 50 mg daily. Study drug (eplerenone) will be paid by the North Florida Foundation for Research and Education for the duration of the study.

   a. Down-titration or termination of non-essential anti-hypertensive agents is permissible so that eplerenone does not result in hypotension. Essential medications are as follows:
   * Angiotensin converting enzyme inhibitors (ACE-inhibitors) or angiotensin receptor blockers, if intolerant to ACE-inhibitors are indicated for treatment left ventricular dysfunction (i.e. left ventricular ejection fraction ≤40%), diabetes, and proteinuric chronic kidney disease.
   * Beta-blockers are indicated 3 years after an acute myocardial infarction, unless there is persistent left ventricular dysfunction (i.e. left ventricular ejection fraction ≤40%).
4. Monitoring.

   a. Serum potassium within the last 30 days is required before initiating eplerenone. Repeat blood draw is required within the first week, and one month after the start of treatment with eplerenone.
5. Quality of life questionnaire. a. The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) will be administered at baseline and 8 weeks. The KCCQ-12 instrument will be mailed to the subject. Study coordinator will call the subject at 8 weeks to confirm vital status, assess if any adverse reactions from eplerenone, and provide assistance to completing the KCCQ-12, if needed.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bavry, MD, Principal Investigator — University of Florida
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at Malcom Randall VA Medical Center
Groups:
- Eplerenone: All subjects will receive eplerenone 50 mg daily. The Kansas City Cardiomyopathy Questionnaire-12 will be administered at baseline and 8 weeks. Serum potassium within the last 30 days is required before initiating eplerenone, repeat blood draw within the first week of starting eplerenone and at 4 weeks.
Period: Overall Study
Arm/Group | Eplerenone
Started | 12
Completed | 8
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — screen failure | 3

BASELINE CHARACTERISTICS:
Population: 12
Groups:
- Eplerenone: All subjects will receive study drug daily.
  Eplerenone: 50mg daily
  Kansas City Cardiomyopathy Questionnaire: administered at baseline and 8 weeks
  Serum potassium: within the last 30 days is required before initiating eplerenone, repeat blood draw within the first week and starting eplerenone and 4 weeks after starting eplerenone
Arm/Group | Eplerenone
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ-12)-Summary Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a self-administered health status survey. The KCCQ-12 has 4 domains (physical limitation, symptom frequency, quality of life, social limitation) and one summary score. Score are scaled 0-100, where 1 denotes the lowest reportable health status and 100 the highest.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Eplerenone: Eplerenone 50 mg daily administered orally to subjects
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
score on a scale
  Baseline | 59.4 (19.7)
  8 weeks | 74.1 (20.0)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.12, t-test, 2 sided

2. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ-12)-Physical Limitation Score
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
score on a scale
  Baseline | 53.0 (21.4)
  8 weeks | 61.5 (14.8)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.49, t-test, 2 sided

3. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ-12)-Symptom Frequency Score
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
score on a scale
  Baseline | 63.5 (20.7)
  8 weeks | 81.5 (14.4)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided

4. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ-12)-Quality of Life Score
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
score on a scale
  Baseline | 54.9 (40.5)
  8 weeks | 73.6 (30.8)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.27, t-test, 2 sided

5. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ-12)-Social Limitation Score
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
score on a scale
  Baseline | 65.6 (32.2)
  8 weeks | 80.1 (26.0)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.18, t-test, 2 sided

6. Secondary Outcome: Systolic Blood Pressure
Description: Cuff systolic blood pressure
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
mm Hg
  Baseline | 122.5 (16.5)
  8 weeks | 120.0 (26.3)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.8, t-test, 2 sided

7. Secondary Outcome: Diastolic Blood Pressure
Description: Cuff diastolic blood pressure
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
mm Hg
  Baseline | 56.2 (7.7)
  8 weeks | 55.0 (6.2)
Statistical Analysis 1: Comparison: Eplerenone; Change from baseline to 8 weeks; Test type: Superiority; p = 0.76, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Eplerenone
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03923530/ICF_000.pdf
  • Study Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03923530/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03923530/SAP_002.pdf